CLINICAL TRIAL: NCT01479621
Title: A 12-Week Dose-ranging Study to Evaluate the Efficacy and Safety of Fluticasone Propionate DPI Administered Twice Daily Compared With Placebo in Adolescent and Adult Subjects With Persistent Asthma Uncontrolled on Non-steroidal Therapy
Brief Title: A Study of the Effectiveness and Safety of Different Doses of Fluticasone Propionate Taken From a Dry Powder Inhaler in Adolescents and Adults Who Have Asthma That is Not Controlled by Asthma Medications Not Containing Steroids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FpS-AS-201; 2010-023600-27 (EudraCT Number)
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Asthma
Keywords: Dose Ranging; Fluticasone Propionate; Dry Powder Inhaler (DPI); Non-steroidal; Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Fp MDPI 12.5 mcg (Experimental): Fluticasone propionate (Fp) 12.5 mcg per dose twice a day (for a total daily dose of 25 mcg) using a multidose dry powder inhaler (MDPI) for 12 weeks in a double-blind manner.
  During the run-in and the treatment periods, all subjects replaced their current rescue medication with albuterol/salbutamol hydrofluoroalkane (HFA) metered dose inhaler (MDI) (90 mcg/actuation) for use on an as needed basis for the relief of asthma symptoms.
  Interventions: Drug: Fp MDPI; Drug: albuterol/salbutamol
- Fp MDPI 25 mcg (Experimental): Fluticasone propionate (Fp) 25 mcg per dose twice a day (for a total daily dose of 50 mcg) using a multidose dry powder inhaler (MDPI) for 12 weeks in a double-blind manner.
  During the run-in and the treatment periods, all subjects replaced their current rescue medication with albuterol/salbutamol hydrofluoroalkane (HFA) metered dose inhaler (MDI) (90 mcg/actuation) for use on an as needed basis for the relief of asthma symptoms.
  Interventions: Drug: Fp MDPI; Drug: albuterol/salbutamol
- Fp MDPI 50 mcg (Experimental): Fluticasone propionate (Fp) 50 mcg per dose twice a day (for a total daily dose of 100 mcg) using a multidose dry powder inhaler (MDPI) for 12 weeks in a double-blind manner.
  During the run-in and the treatment periods, all subjects replaced their current rescue medication with albuterol/salbutamol hydrofluoroalkane (HFA) metered dose inhaler (MDI) (90 mcg/actuation) for use on an as needed basis for the relief of asthma symptoms.
  Interventions: Drug: Fp MDPI; Drug: albuterol/salbutamol
- Fp MDPI 100 mcg (Experimental): Fluticasone propionate (Fp) 100 mcg per dose twice a day (for a total daily dose of 200 mcg) using a multidose dry powder inhaler (MDPI) for 12 weeks in a double-blind manner.
  During the run-in and the treatment periods, all subjects replaced their current rescue medication with albuterol/salbutamol hydrofluoroalkane (HFA) metered dose inhaler (MDI) (90 mcg/actuation) for use on an as needed basis for the relief of asthma symptoms.
  Interventions: Drug: Fp MDPI; Drug: albuterol/salbutamol
- Placebo MDPI (Experimental): Placebo twice a day using a multidose dry powder inhaler (MDPI) for 12 weeks in a double-blind manner. During the run-in and the treatment periods, all subjects replaced their current rescue medication with albuterol/salbutamol hydrofluoroalkane (HFA) metered dose inhaler (MDI) (90 mcg/actuation) for use on an as needed basis for the relief of asthma symptoms.
  Interventions: Drug: albuterol/salbutamol; Drug: Placebo MDPI
- Flovent Diskus 100mcg (Experimental): Fluticasone propionate (Fp) 100 mcg per dose twice a day (for a total daily dose of 200 mcg) using a multidose dry powder inhaler (MDPI) for 12 weeks in an open-label manner.
  During the run-in and the treatment periods, all subjects replaced their current rescue medication with albuterol/salbutamol hydrofluoroalkane (HFA) metered dose inhaler (MDI) (90 mcg/actuation) for use on an as needed basis for the relief of asthma symptoms.
  Interventions: Drug: Flovent Diskus; Drug: albuterol/salbutamol

INTERVENTIONS:
Drug: Fp MDPI — Fp MDPI is an inhalation-driven multidose dry powder inhaler (MDPI) containing fluticasone propionate (Fp) dispersed in a lactose monohydrate excipient and contained within a reservoir. A metered dose of drug is delivered to a dose cup via an air pulse activated when the cap is opened.
  During the treatment period, participants were randomized to 12.5, 25, 50 or 100 mcg of Fp one inhalation twice a day for a total daily dose of 25, 50, 100 or 200 mcg. Study drug was administered in the morning and in the evening
  Other Names: Fluticasone propionate; Fp SPIROMAX® Inhalation Powder
  Arms: Fp MDPI 100 mcg; Fp MDPI 12.5 mcg; Fp MDPI 25 mcg; Fp MDPI 50 mcg
Drug: Flovent Diskus — Flovent Diskus contains the active ingredient fluticasone propionate (Fp). Flovent Diskus 100 mcg was used twice a day, once in the morning and evening, for a total daily dose of 200 mcg of Fp. This therapy was not blinded as the inhaler device was different than the MDPI used in the other treatment arms.
  Other Names: Fluticasone propionate
  Arms: Flovent Diskus 100mcg
Drug: albuterol/salbutamol — A short-acting β2-adrenergic agonists (SABA), albuterol/salbutamol hydrofluoroalkane (HFA) metered dose inhaler (MDI), was provided to be used as needed for the relief of asthma symptoms during both the run-in and treatment periods (to replace the subject's current rescue medication).
  Other Names: short-acting β2-adrenergic agonists
Drug: Placebo MDPI — Placebo multidose dry powder inhaler in the morning and evening. Placebo MDPI was provided in devices identical in appearance to Fp MDPI.
  Arms: Placebo MDPI

SUMMARY:
This is a randomized, double-blind, placebo- and open-label active controlled, parallel-group, multicenter, dose ranging study in male or female subjects ages 12 years and older with persistent asthma who are uncontrolled on non-steroidal therapy. The primary objective of this study is to evaluate the dose response, efficacy and safety of 4 different doses of fluticasone propionate delivered as Fluticasone Propionate DPI (Dry Powder Inhaler) when administered twice daily.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent/assent signed and dated by the subject and/or parent /legal guardian before conducting any study related procedure.
2. Male or female 12 years and older, as of the Screening Visit. Male or female 18 years and older, as of the Screening Visit, in countries where local regulations or the regulatory status of study medication permit enrollment of adults only.
3. General good health, and free of any concomitant conditions or treatment that could interfere with study conduct, influence the interpretation of study observations/results, or put the subject at increased risk during the study.
4. Asthma Diagnosis: Asthma as defined by the National Institutes of Health (NIH).
5. Severity of Disease: A best forced expiratory volume in one second (FEV1) of 40%-85% of the predicted normal value during the Screening Visit. NHANES III predicted values will be used for subjects aged ≥12 years and adjustments to predicted values will be made for African American subjects.
6. Reversibility of Disease: Demonstrated a ≥15% reversibility of FEV1 within 30 minutes following 2 inhalations of albuterol/salbutamol inhalation aerosol (if required, spacers are permitted for reversibility testing only) at the Screening Visit. If a subject fails to demonstrate an increase in FEV1 ≥15%, then the subject is not eligible for the study and will not be allowed to re-screen.
7. Current Asthma Therapy: Subjects must be on a short-acting β2-agonist alone or a non-corticosteroid maintenance medication (with or without a short-acting β2-agonist) for ≥ 3 months preceding the Screening Visit. Subjects must not have used an inhaled corticosteroid for at least 6 weeks preceding the Screening Visit.

   Exception: Based upon the investigator's judgment that there is no inherent harm in changing the subject's current ICS therapy and the subject provides consent, subjects on low dose ICS (100mcg Fp BID or equivalent) may be switched to a short-acting β2 agonist alone at a Pre-screening Visit. The subject will be required to return to the clinic to complete the Screening Visit once the 2-week washout period has been completed.
8. Short-Acting β2-Agonists: All subjects must be able to replace their current short-acting β2-agonists with albuterol/salbutamol inhalation aerosol at the Screening Visit for use as needed for the duration of the study. The use of spacer devices with the metered dose inhaler (MDI) will not be allowed during the study with exception of its use during reversibility testing at the Screening Visit. Nebulized albuterol/salbutamol will not be allowed at any time during the study. Subjects must be able to withhold all inhaled short-acting beta sympathomimetic bronchodilators for at least 6 hours prior to all study visits.
9. If female, is currently not pregnant, breast feeding, or attempting to become pregnant, has a negative serum pregnancy test, and is of

   1. Non-childbearing potential, defined as:

      * Before menarche or > or =1 year post-menopausal or
      * Surgically sterile (tubal ligation, bilateral oophorectomy, or hysterectomy) or
      * Congenital sterility or
      * Diagnosed as infertile and not undergoing treatment to reverse infertility or is of
   2. Child-bearing potential, willing to commit to using a consistent and acceptable method of birth control as defined below for the duration of the study:

      * Systemic contraception used for > or = 1 month prior to screening, including birth control pills, transdermal patch (Ortho Evra®), vaginal ring (NuvaRing®), levonorgesterel (Norplant®), or injectable progesterone (Depo-Provera®) or
      * Double barrier methods (condoms, cervical cap, diaphragm, and vaginal contraceptive film with spermicide) or
      * Intrauterine device (IUD) or is of
   3. Child-bearing potential and not sexually active, willing to commit to using a consistent and acceptable method of birth control as defined above for the duration of the study, in the event the subject becomes sexually active.
10. Capable of understanding the requirements, risks, and benefits of study participation, and, as judged by the investigator, capable of giving informed consent/assent and being compliant with all study requirements (visits, record-keeping, etc).

Exclusion Criteria:

1. History of life-threatening asthma that is defined for this protocol as an asthma episode that required intubation and/or was associated with hypercapnea, respiratory arrest or hypoxic seizures.
2. Culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus, or middle ear that is not resolved within 2 weeks prior to the Screening Visit. In addition, the subject must be excluded if such infection occurs between the Screening Visit and the Randomization Visit.
3. Any asthma exacerbation requiring oral corticosteroids within 3 months of the Screening Visit. A subject must not have had any hospitalization for asthma within 6 months prior to the Screening Visit.

   Note: An exacerbation of asthma is defined as any worsening of asthma requiring any treatment other than rescue albuterol/salbutamol HFA MDI and/or the subject's regular non-corticosteroid maintenance treatment. This includes requiring the use of systemic corticosteroids and/or emergency room visit or hospitalization, a change in the subject's regular non-corticosteroid maintenance treatment, or the addition of other asthma medications.
4. Presence of glaucoma, cataracts, ocular herpes simplex, or malignancy other than basal cell carcinoma.
5. Historical or current evidence of a clinically significant disease including, but not limited to: cardiovascular (e.g., congestive heart failure, known aortic aneurysm, clinically significant cardiac arrhythmia or coronary heart disease), hepatic, renal, hematological, neuropsychological, endocrine (e.g., uncontrolled diabetes mellitus, uncontrolled thyroid disorder, Addison's disease, Cushing's syndrome), gastrointestinal (e.g., poorly-controlled peptic ulcer, GERD), or pulmonary (e.g., chronic bronchitis, emphysema, bronchiectasis with the need for treatment, cystic fibrosis, bronchopulmonary dysplasia, chronic obstructive pulmonary disease). Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which could affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
6. Have any of the following conditions that, in the judgment of the investigator, might cause participation in this study to be detrimental to the subject, including, but not limited to:

   * Current malignancy excluding basal cell carcinoma; History of malignancy is acceptable only if the subject has been in remission for one year prior to the Screening Visit. (Remission is defined as no current evidence of malignancy and no treatment for the malignancy in the 12 months prior to the Screening Visit)
   * Current or untreated tuberculosis; History of tuberculosis is acceptable only if a subject has received an approved prophylactic treatment regimen or an approved active treatment regimen and has had no evidence of active disease for a minimum of 2 years • Uncontrolled hypertension (systolic BP ≥160 or diastolic BP >100)
   * Stroke within 3 months prior to the Screening Visit
   * Immunologic compromise
7. History of a positive test for HIV, hepatitis B or hepatitis C infection.
8. Clinical visual evidence of oral candidiasis at the Screening Visit.
9. History of any adverse reaction, including immediate or delayed hypersensitivity to any β2-agonist, sympathomimetic drug, or any intranasal, inhaled, or systemic corticosteroid therapy. Known or suspected sensitivity to the constituents of the dry powder inhalers (Spiromax or Diskus) used in the study (i.e., lactose).
10. History of severe allergy to milk protein.
11. Use of systemic, oral or depot corticosteroids within 12 weeks prior to the Screening Visit

    * Use of topical corticosteroids (≤1% hydrocortisone cream) for dermatological disease is permitted
    * Use of intranasal corticosteroids at a stable dose for at least 4 weeks prior to the Screening Visit and throughout the study is permitted
12. Use of immunosuppressive medications within 4 weeks prior to the Screening Visit and during the study.
13. Immunotherapy at a stable dose for at least 90 days prior to the Screening Visit and throughout the study for the treatment of allergies is permitted.
14. Use of potent Cytochrome P450 3A4 (CYP3A4) inhibitors (e.g., ritonavir, ketoconazole, itraconazole) within 4 weeks prior to the Screening Visit.
15. History of alcohol or drug abuse within two years preceding the Screening Visit.
16. Current smoker or a smoking history of 10 pack years or more (a pack year is defined as smoking 1 pack of cigarettes/day for 1 year). A subject may not have used tobacco products within the past one year (e.g., cigarettes, cigars, chewing tobacco, or pipe tobacco).
17. Study participation by clinical investigator site employees and/or their immediate relatives.
18. Study participation by more than one subject from the same household at the same time. However, after the study completion or discontinuation by one subject another subject from the same household may be screened.
19. Participation in any investigational drug study within the 30 days (starting at the final follow-up visit) preceding the Screening Visit or planned participation in another investigational drug study at any time during this study.
20. Pregnancy, nursing, or plans to become pregnant or donate gametes (ova or sperm) for in vitro fertilization during the study period or for 30 days following the subject's last study related visit (for eligible subjects only - if applicable). Eligible female subjects unwilling to employ appropriate contraceptive measures to ensure that pregnancy will not occur during the study will be excluded.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 909 (Actual)
Dates: Start 2012-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (189):
- United States (129):
  - Teva Investigational Site 10165, Homewood, Alabama
  - Teva Investigational Site 11142, Goodyear, Arizona
  - Teva Investigational Site 10104, Scottsdale, Arizona
  - Teva Investigational Site 11149, Little Rock, Arkansas
  - Teva Investigational Site 10173, Bakersfield, California
  - Teva Investigational Site 10163, Costa Mesa, California
  - Teva Investigational Site 10156, Encinitas, California
  - Teva Investigational Site 11101, Fountain Valley, California
  - Teva Investigational Site 11111, Fresno, California
  - Teva Investigational Site 10151, Granada Hills, California
  - Teva Investigational Site 10157, Huntington Beach, California
  - Teva Investigational Site 10176, Huntington Beach, California
  - Teva Investigational Site 10147, Long Beach, California
  - Teva Investigational Site 11110, Napa, California
  - Teva Investigational Site 10136, Newport Beach, California
  - Teva Investigational Site 11122, North Hollywood, California
  - Teva Investigational Site 10140, Orange, California
  - Teva Investigational Site 10197, Palmdale, California
  - Teva Investigational Site 10185, Redwood City, California
  - Teva Investigational Site 10143, Riverside, California
  - Teva Investigational Site 11137, Roseville, California
  - Teva Investigational Site 10130, San Diego, California
  - Teva Investigational Site 10182, San Diego, California
  - Teva Investigational Site 10179, San Jose, California
  - Teva Investigational Site 10106, Stockton, California
  - Teva Investigational Site 10129, Walnut Creek, California
  - Teva Investigational Site 10145, Centennial, Colorado
  - Teva Investigational Site 10172, Colorado Springs, Colorado
  - Teva Investigational Site 10133, Denver, Colorado
  - Teva Investigational Site 10154, Denver, Colorado
  - Teva Investigational Site 11146, Denver, Colorado
  - Teva Investigational Site 10128, Wheat Ridge, Colorado
  - Teva Investigational Site 10196, Waterbury, Connecticut
  - Teva Investigational Site 10191, Boynton Beach, Florida
  - Teva Investigational Site 11127, Brandon, Florida
  - Teva Investigational Site 11118, Clearwater, Florida
  - Teva Investigational Site 11141, Hialeah, Florida
  - Teva Investigational Site 11140, Kissimmee, Florida
  - Teva Investigational Site 10137, Miami, Florida
  - Teva Investigational Site 10153, Miami, Florida
  - Teva Investigational Site 11120, Miami, Florida
  - Teva Investigational Site 11128, Miami, Florida
  - Teva Investigational Site 11132, Miami, Florida
  - Teva Investigational Site 11145, Miami, Florida
  - Teva Investigational Site 10171, Ocala, Florida
  - Teva Investigational Site 10178, Sarasota, Florida
  - Teva Investigational Site 11103, South Miami, Florida
  - Teva Investigational Site 10161, Tallahassee, Florida
  - Teva Investigational Site 10139, Tampa, Florida
  - Teva Investigational Site 11114, Albany, Georgia
  - Teva Investigational Site 10111, Columbus, Georgia
  - Teva Investigational Site 11124, Columbus, Georgia
  - Teva Investigational Site 10180, Gainesville, Georgia
  - Teva Investigational Site 10168, Lawrenceville, Georgia
  - Teva Investigational Site 11109, Idaho Falls, Idaho
  - Teva Investigational Site 10116, Meridian, Idaho
  - Teva Investigational Site 10127, South Bend, Indiana
  - Teva Investigational Site 10184, Iowa City, Iowa
  - Teva Investigational Site 10113, Metairie, Louisiana
  - Teva Investigational Site 10164, Bangor, Maine
  - Teva Investigational Site 10158, Bethesda, Maryland
  - Teva Investigational Site 10110, Largo, Maryland
  - Teva Investigational Site 10177, Wheaton, Maryland
  - Teva Investigational Site 10138, North Dartmouth, Massachusetts
  - Teva Investigational Site 10146, North Dartmouth, Massachusetts
  - Teva Investigational Site 10131, Minneapolis, Minnesota
  - Teva Investigational Site 10175, St Louis, Missouri
  - Teva Investigational Site 10189, St Louis, Missouri
  - Teva Investigational Site 11147, St Louis, Missouri
  - Teva Investigational Site 10118, Bellevue, Nebraska
  - Teva Investigational Site 10150, Omaha, Nebraska
  - Teva Investigational Site 11144, Omaha, Nebraska
  - Teva Investigational Site 11136, Henderson, Nevada
  - Teva Investigational Site 10114, Brick, New Jersey
  - Teva Investigational Site 10193, Cherry Hill, New Jersey
  - Teva Investigational Site 10101, Hillsborough, New Jersey
  - Teva Investigational Site 10155, Skillman, New Jersey
  - Teva Investigational Site 10188, West Orange, New Jersey
  - Teva Investigational Site 11113, Albuquerque, New Mexico
  - Teva Investigational Site 10187, Brooklyn, New York
  - Teva Investigational Site 10120, New York, New York
  - Teva Investigational Site 10190, Newburgh, New York
  - Teva Investigational Site 10167, North Syracuse, New York
  - Teva Investigational Site 10112, Rochester, New York
  - Teva Investigational Site 10105, High Point, North Carolina
  - Teva Investigational Site 10122, Raleigh, North Carolina
  - Teva Investigational Site 10194, Canton, Ohio
  - Teva Investigational Site 10107, Cincinnati, Ohio
  - Teva Investigational Site 10123, Cincinnati, Ohio
  - Teva Investigational Site 10144, Columbus, Ohio
  - Teva Investigational Site 11135, Dayton, Ohio
  - Teva Investigational Site 11115, Middleburg Heights, Ohio
  - Teva Investigational Site 10160, Oklahoma City, Oklahoma
  - Teva Investigational Site 10174, Oklahoma City, Oklahoma
  - Teva Investigational Site 10198, Oklahoma City, Oklahoma
  - Teva Investigational Site 11108, Ashland, Oregon
  - Teva Investigational Site 10132, Eugene, Oregon
  - Teva Investigational Site 10135, Medford, Oregon
  - Teva Investigational Site 10142, Portland, Oregon
  - Teva Investigational Site 11104, Normal Square, Pennsylvania
  - Teva Investigational Site 10183, Philadelphia, Pennsylvania
  - Teva Investigational Site 10166, Pittsburgh, Pennsylvania
  - Teva Investigational Site 10121, Upland, Pennsylvania
  - Teva Investigational Site 11119, East Providence, Rhode Island
  - Teva Investigational Site 10181, Lincoln, Rhode Island
  - Teva Investigational Site 10162, Providence, Rhode Island
  - Teva Investigational Site 10126, Charleston, South Carolina
  - Teva Investigational Site 10149, Charleston, South Carolina
  - Teva Investigational Site 10199, Orangeburg, South Carolina
  - Teva Investigational Site 11131, Spartanburg, South Carolina
  - Teva Investigational Site 10119, Boerne, Texas
  - Teva Investigational Site 10141, Dallas, Texas
  - Teva Investigational Site 10192, Dallas, Texas
  - Teva Investigational Site 10148, El Paso, Texas
  - Teva Investigational Site 10115, San Antonio, Texas
  - Teva Investigational Site 11133, San Antonio, Texas
  - Teva Investigational Site 11134, San Antonio, Texas
  - Teva Investigational Site 10103, Waco, Texas
  - Teva Investigational Site 11143, Layton, Utah
  - Teva Investigational Site 10195, Provo, Utah
  - Teva Investigational Site 10134, South Burlington, Vermont
  - Teva Investigational Site 10159, Burke, Virginia
  - Teva Investigational Site 10102, Fairfax, Virginia
  - Teva Investigational Site 11105, Manassas, Virginia
  - Teva Investigational Site 10108, Richmond, Virginia
  - Teva Investigational Site 10124, Spokane, Washington
  - Teva Investigational Site 11117, Tacoma, Washington
  - Teva Investigational Site 11125, Tacoma, Washington
  - Teva Investigational Site 10170, Greenfield, Wisconsin
- Bulgaria (7):
  - Teva Investigational Site 59107, Burgas
  - Teva Investigational Site 59103, Lovech
  - Teva Investigational Site 59106, Pleven
  - Teva Investigational Site 59104, Rousse
  - Teva Investigational Site 59101, Sofia
  - Teva Investigational Site 59102, Sofia
  - Teva Investigational Site 59105, Sofia
- Croatia (4):
  - Teva Investigational Site 85105, Split
  - Teva Investigational Site 85102, Zagreb
  - Teva Investigational Site 85103, Zagreb
  - Teva Investigational Site 85104, Zagreb
- Hungary (11):
  - Teva Investigational Site 36107, Balassagyarmat
  - Teva Investigational Site 36104, Budapest
  - Teva Investigational Site 36105, Budapest
  - Teva Investigational Site 36113, Csoma
  - Teva Investigational Site 36103, Miskolc
  - Teva Investigational Site 36108, Mosdós
  - Teva Investigational Site 36102, Nyíregyháza
  - Teva Investigational Site 36106, Szeged
  - Teva Investigational Site 36109, Szeged
  - Teva Investigational Site 36101, Szombathely
  - Teva Investigational Site 36111, Tatabánya
- Israel (10):
  - Teva Investigational Site 72111, Ashkelon
  - Teva Investigational Site 72101, Haifa
  - Teva Investigational Site 72102, Jerusalem
  - Teva Investigational Site 72104, Jerusalem
  - Teva Investigational Site 72109, Kfar Saba
  - Teva Investigational Site 72106, Petah Tikva
  - Teva Investigational Site 72107, Ramat Gan
  - Teva Investigational Site 72103, Rehovot
  - Teva Investigational Site 72108, Tel Aviv
  - Teva Investigational Site 72110, Tel Aviv
- Poland (7):
  - Teva Investigational Site 48107, Bialystok
  - Teva Investigational Site 48105, Bydgoszcz
  - Teva Investigational Site 48106, Grodzisk Mazowiecki
  - Teva Investigational Site 48101, Lodz
  - Teva Investigational Site 48108, Poznan
  - Teva Investigational Site 48103, Tarnów
  - Teva Investigational Site 48104, Wroclaw
- Serbia (2):
  - Teva Investigational Site 81101, Belgrade
  - Teva Investigational Site 81102, Belgrade
- Spain (3):
  - Teva Investigational Site 34101, Badalona
  - Teva Investigational Site 34102, Barcelona
  - Teva Investigational Site 34103, Salt
- Ukraine (16):
  - Teva Investigational Site 80101, Dnipropetrovsk
  - Teva Investigational Site 80113, Dnipropetrovsk
  - Teva Investigational Site 80111, Donetsk
  - Teva Investigational Site 80103, Kharkiv
  - Teva Investigational Site 80117, Kharkiv
  - Teva Investigational Site 80104, Kyiv
  - Teva Investigational Site 80105, Kyiv
  - Teva Investigational Site 80106, Kyiv
  - Teva Investigational Site 80107, Kyiv
  - Teva Investigational Site 80108, Kyiv
  - Teva Investigational Site 80109, Kyiv
  - Teva Investigational Site 80114, Odesa
  - Teva Investigational Site 80118, Ternopil
  - Teva Investigational Site 80112, Vinnytsia
  - Teva Investigational Site 80115, Yalta
  - Teva Investigational Site 80110, Zaporizhzhia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1903 subjects with asthma were screened for enrollment into this study. Of the 994 subjects who were not enrolled, 983 were excluded on the basis of inclusion/exclusion criteria and 6 subjects withdrew consent, and for 5 the reason given was "other".
Pre-assignment Details: 909 subjects at 188 centers met entry criteria and were considered to be eligible for enrollment into the run-in period of the study.
Groups:
- Placebo MDPI (Run-In): Upon enrollment, participants used current asthma medications and 1 inhalation of placebo multidose dry powder inhaler (MDPI), single-blind, twice daily for 14-day (±2 days).
Period: Pre-Assignment Period (Run-In Placebo)
Arm/Group | Placebo MDPI (Run-In) | Fp MDPI 12.5 mcg | Fp MDPI 25 mcg | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Placebo MDPI | Flovent Diskus 100mcg
Started | 909 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 622 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 287 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Inclusion/exclusion criteria | 93 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 19 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Randomization criteria not met | 153 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 7 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 15 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period
Arm/Group | Placebo MDPI (Run-In) | Fp MDPI 12.5 mcg | Fp MDPI 25 mcg | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Placebo MDPI | Flovent Diskus 100mcg
Started | 0 | 103 | 104 | 104 | 103 | 104 | 104
Safety Population | 0 | 103 | 104 | 104 | 103 | 104 | 104
Full Analysis Set | 0 | 102 | 101 | 102 | 102 | 102 | 102
Completed | 0 | 79 | 83 | 92 | 82 | 63 | 84
Not Completed | 0 | 24 | 21 | 12 | 21 | 41 | 20
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 4 | 2 | 2 | 5 | 5 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Non-compliance to study drug | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 9 | 6 | 5 | 2 | 10 | 6
Not completed — Pregnancy | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Sponsor request subject to be withdrawn | 0 | 2 | 3 | 1 | 1 | 1 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 2 | 2 | 1
Not completed — Met stopping criteria | 0 | 8 | 7 | 4 | 9 | 20 | 6

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | Fp MDPI 12.5 mcg | Fp MDPI 25 mcg | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Placebo MDPI | Flovent Diskus 100mcg | Total
Number analyzed (Participants) | 103 | 104 | 104 | 103 | 104 | 104 | 622
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (16.94) | 42.4 (16.02) | 39.1 (16.06) | 36.9 (15.34) | 39.7 (15.28) | 40.0 (15.34) | 39.9 (15.87)
Age, Customized [Count of Participants; unit: Participants]
  12-17 years | 10 | 7 | 14 | 9 | 5 | 7 | 52
  Adults (18-64 years) | 85 | 90 | 86 | 88 | 93 | 93 | 535
  Adults (65+ years) | 8 | 7 | 4 | 6 | 6 | 4 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 63 | 60 | 60 | 55 | 63 | 358
  Male | 46 | 41 | 44 | 43 | 49 | 41 | 264
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 91 | 91 | 90 | 85 | 85 | 85 | 527
  Black | 10 | 11 | 12 | 14 | 17 | 17 | 81
  Asian | 1 | 2 | 2 | 4 | 0 | 1 | 10
  American Indian or Alaskan Native | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Other | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 4 | 7 | 13 | 11 | 6 | 50
  Not Hispanic or Latino | 94 | 100 | 97 | 90 | 93 | 98 | 572
Weight [Mean (Standard Deviation); unit: kg] | 82.0 (23.29) | 80.4 (19.62) | 78.7 (23.08) | 84.6 (23.51) | 80.5 (20.00) | 81.5 (23.53) | 81.3 (22.22)
Height [Mean (Standard Deviation); unit: cm] | 168.8 (10.54) | 169.2 (8.89) | 168.6 (10.33) | 168.7 (10.94) | 169.5 (9.25) | 169.0 (9.39) | 169.0 (9.88)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.7 (7.43) | 28.1 (6.47) | 27.5 (6.78) | 29.6 (7.54) | 28.0 (6.61) | 28.4 (7.31) | 28.4 (7.04)
Forced Expiratory Volume in 1 Second (FEV1) [Mean (Standard Deviation); unit: liters] | 2.3 (0.69) | 2.2 (0.59) | 2.2 (0.63) | 2.3 (0.66) | 2.3 (0.62) | 2.2 (0.66) | 2.2 (0.64)
% Predicted Expiratory Volume In 1 Second [Mean (Standard Deviation); unit: percent predicted FEV1] | 66.6 (11.80) | 67.5 (10.50) | 66.3 (11.15) | 66.4 (11.61) | 66.4 (11.14) | 65.3 (11.74) | 66.4 (11.30)
Qualifying Airway Reversibility [Mean (Standard Deviation); unit: percentage increase in FEV1] — Patients demonstrated a ≥15% reversibility of FEV1 within 30 minutes following 2-4 inhalations of albuterol/salbutamol inhalation aerosol at the screening visit. If subjects failed to demonstrate an increase in FEV1 ≥15% then subjects were not eligible for the study; however, based on investigator judgment, they were allowed to retest once within 7 days. Reversibility values of 14.50 through 14.99% were rounded to 15%.
  percentage increase in FEV1 | 26.7 (12.01) | 26.0 (11.86) | 24.3 (10.63) | 27.6 (12.92) | 30.6 (17.84) | 26.2 (12.50) | 26.9 (13.25)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline In Trough (Morning Predose And Pre-Rescue Bronchodilator) Forced Expiratory Volume In 1 Second (FEV1) Over The 12-Week Treatment Period
Description: Trough FEV1 was measured electronically by spirometry at morning (AM) investigational site visits, before administration of the AM dose of study drug and before albuterol/salbutamol administration. The highest FEV1 value from 3 acceptable and 2 reproducible maneuvers was used. All FEV1 data were submitted to a central reading center for evaluation.
  The p-values for the treatment comparisons to placebo are from an MMRM model excluding FLOVENT DISKUS data: change from baseline = baseline FEV1 + sex + age + treatment + visit + treatment*visit with an unstructured covariance matrix assumed.
Time Frame: Baseline (Day 1, pre-dose), During Study (Days 7, 14, 28, 56 and 84 pre-dose)
Population: Full analysis set, (participants who contributed >=1 to the analysis). Data from one site omitted due to GCP concerns. Flovent Diskus data was used for confirmatory and exploratory endpoints (see outcome #11).
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Fp MDPI 12.5 mcg | Fp MDPI 25 mcg | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Placebo MDPI | Flovent Diskus 100mcg
Number analyzed (Participants) | 94 | 97 | 100 | 94 | 94 | 0
liters | 0.170 (0.0300) | 0.229 (0.0295) | 0.243 (0.0288) | 0.267 (0.0300) | 0.118 (0.0302) |
Statistical Analysis 1: Comparison: Fp MDPI 12.5 mcg vs Fp MDPI 25 mcg vs Fp MDPI 50 mcg vs Fp MDPI 100 mcg vs Placebo MDPI; A linear in log-dose trend contrast evaluated the time-averaged dose-response trend, where the logarithm of dose was defined as log(dose+1) to accommodate the case of a zero dose (placebo). A fixed-sequence testing procedure was employed to control the overall Type I error rate at the 0.05 level. Specifically, the 2-sided linear in log-dose time-averaged trend test was first performed followed by pairwise comparisons of each Fp MDPI dose versus placebo; Test type: Superiority or Other; p = 0.0001, Regression, Linear — The study was considered positive if the trend test was positive and the test involving the highest Fp MDPI dose (100 mcg twice daily) indicated significantly greater time averaged FEV1 mean than placebo
Statistical Analysis 2: Comparison: Fp MDPI 100 mcg vs Placebo MDPI; This is the second analysis in the fixed-sequence testing procedure employed to control the overall Type I error rate at the 0.05 level; Test type: Superiority or Other; p = 0.0005, mixed model for repeated measures — [p-value comment as in outcome 1, analysis 1]; LSM difference = 0.149, 95% CI 2-sided [0.066 to 0.233]
Statistical Analysis 3: Comparison: Fp MDPI 50 mcg vs Placebo MDPI; This is the third analysis in the fixed-sequence testing procedure employed to control the overall Type I error rate at the 0.05 level; Test type: Superiority or Other; p = 0.0027, mixed model for repeated measures; LSM difference = 0.126, 95% CI 2-sided [0.044 to 0.208]
Statistical Analysis 4: Comparison: Fp MDPI 25 mcg vs Placebo MDPI; This is the fourth analysis in the fixed-sequence testing procedure employed to control the overall Type I error rate at the 0.05 level; Test type: Superiority or Other; p = 0.0086, mixed model for repeated measures; LSM difference = 0.111, 95% CI 2-sided [0.028 to 0.194]
Statistical Analysis 5: Comparison: Fp MDPI 12.5 mcg vs Placebo MDPI; This is the fifth analysis in the fixed-sequence testing procedure employed to control the overall Type I error rate at the 0.05 level; Test type: Superiority or Other; p = 0.2227, mixed model for repeated measures; LSM difference = 0.052, 95% CI 2-sided [-0.032 to 0.136]

2. Secondary Outcome: Change From Baseline In Weekly Average Of Daily Trough (Predose And Pre-Rescue Bronchodilator) Morning Peak Expiratory Flow (PEF) Over The 12-Week Treatment Period
Description: Peak expiratory flow was determined in the AM and in the PM, before administration of study or rescue medications using a handheld electronic peak flow meter. The highest value of triplicate measurements obtained was recorded by the subject's diary device.
  On mornings for which a treatment visit was scheduled (TV1 through TV9), the PEF was measured and recorded at the investigational site visit.
  Baseline trough AM PEF was defined as the average of recorded (non-missing) trough AM PEF assessments over the 7 days directly preceding first study drug intake.
  The p-values for the treatment comparisons to placebo are from an MMRM model excluding FLOVENT DISKUS data: change from baseline = baseline PEF + sex + age + treatment + visit + treatment*visit with an unstructured covariance matrix assumed.
Time Frame: Baseline (Days -7 to 1, am pre-dose), During Study (Days 2-84 am pre-dose)
Population: Full analysis set, (participants who contributed >=1 to the analysis). Data from one site omitted due to GCP concerns. Flovent Diskus data was used for confirmatory and exploratory endpoints (see outcome #12).
Measure: Least Squares Mean (Standard Error); unit: liters/minute
Arm/Group | Fp MDPI 12.5 mcg | Fp MDPI 25 mcg | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Placebo MDPI | Flovent Diskus 100mcg
Number analyzed (Participants) | 94 | 97 | 99 | 94 | 92 | 0
liters/minute | 30.99 (4.600) | 21.01 (4.521) | 29.58 (4.396) | 27.55 (4.610) | 9.26 (4.755) |
Statistical Analysis 1: Comparison: Fp MDPI 12.5 mcg vs Fp MDPI 25 mcg vs Fp MDPI 50 mcg vs Fp MDPI 100 mcg vs Placebo MDPI; A linear in log-dose trend contrast evaluated the time-averaged dose-response trend, where the logarithm of dose was defined as log(dose+1) to accommodate the case of a zero dose (placebo); Test type: Superiority or Other; p = 0.0017, Regression, Linear — Significance at 0.05
Statistical Analysis 2: Comparison: Fp MDPI 100 mcg vs Placebo MDPI; Test type: Superiority or Other; p = 0.0060, mixed model for repeated measures — Significance at 0.05; LSM difference = 18.29, 95% CI 2-sided [5.28 to 31.29]
Statistical Analysis 3: Comparison: Fp MDPI 50 mcg vs Placebo MDPI; Test type: Superiority or Other; p = 0.0018, mixed model for repeated measures — Significance at 0.05; LSM difference = 20.32, 95% CI 2-sided [7.61 to 33.03]
Statistical Analysis 4: Comparison: Fp MDPI 25 mcg vs Placebo MDPI; Test type: Superiority or Other; p = 0.0741, mixed model for repeated measures — Significance at 0.05; LSM difference = 11.75, 95% CI 2-sided [-1.15 to 24.64]
Statistical Analysis 5: Comparison: Fp MDPI 12.5 mcg vs Placebo MDPI; Test type: Superiority or Other; p = 0.0011, mixed model for repeated measures — Significance at 0.05; LSM difference = 21.72, 95% CI 2-sided [8.73 to 34.72]

3. Secondary Outcome: Change From Baseline In Weekly Average Of Daily Evening Peak Expiratory Flow (PEF) Over The 12-Week Treatment Period
Description: Peak expiratory flow was determined in the AM and in the PM, before administration of study or rescue medications using a handheld electronic peak flow meter. The highest value of triplicate measurements obtained was recorded by the subject's diary device.
  PM PEF baseline was defined as the average of recorded (nonmissing) PM PEF assessments over the 7 days directly preceding first study drug intake.
  The p-values for the treatment comparisons to placebo are from an MMRM model excluding FLOVENT DISKUS data: change from baseline = baseline PEF + sex + age + treatment + visit + treatment*visit with an unstructured covariance matrix assumed.
Time Frame: Baseline (Days -7 to 1, am pre-dose), During Study (Days 2-84 am pre-dose)
Population: Full analysis set, (participants who contributed >=1 to the analysis). Data from one site omitted due to GCP concerns. Flovent Diskus data was used for confirmatory and exploratory endpoints (see outcome #13).
Measure: Least Squares Mean (Standard Error); unit: liters/minute
Arm/Group | Fp MDPI 12.5 mcg | Fp MDPI 25 mcg | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Placebo MDPI | Flovent Diskus 100mcg
Number analyzed (Participants) | 92 | 98 | 99 | 92 | 92 | 0
liters/minute | 27.65 (4.474) | 18.69 (4.347) | 22.20 (4.237) | 20.48 (4.490) | 9.42 (4.588) |
Statistical Analysis 1: Comparison: Fp MDPI 12.5 mcg vs Fp MDPI 25 mcg vs Fp MDPI 50 mcg vs Fp MDPI 100 mcg vs Placebo MDPI; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0434, Regression, Linear — Significance at 0.05
Statistical Analysis 2: Comparison: Fp MDPI 100 mcg vs Placebo MDPI; Test type: Superiority or Other; p = 0.0852, mixed model for repeated measures — Significance at 0.05; LSM difference = 11.06, 95% CI 2-sided [-1.54 to 23.66]
Statistical Analysis 3: Comparison: Fp MDPI 50 mcg vs Placebo MDPI; Test type: Superiority or Other; p = 0.0411, mixed model for repeated measures — Significance at 0.05; LSM difference = 12.78, 95% CI 2-sided [0.52 to 25.04]
Statistical Analysis 4: Comparison: Fp MDPI 25 mcg vs Placebo MDPI; Test type: Superiority or Other; p = 0.1428, mixed model for repeated measures — Significance at 0.05; LSM difference = 9.28, 95% CI 2-sided [-3.14 to 21.69]
Statistical Analysis 5: Comparison: Fp MDPI 12.5 mcg vs Placebo MDPI; Test type: Superiority or Other; p = 0.0046, mixed model for repeated measures — Significance at 0.05; LSM difference = 18.23, 95% CI 2-sided [5.64 to 30.82]

4. Secondary Outcome: Change From Baseline in the Percentage of Rescue-Free 24-hour Periods During the 12-Week Treatment Period
Description: The number of inhalations of rescue medication used each day and each night was recorded in the subject's diary device.
  Change from baseline in the percentage of rescue-free 24-hour periods was analyzed with a marginal (also called population averaged) logistic model. The model included 2 time points of measurement for each subject: the baseline and the treatment period. The model contained covariates for sex, age, and treatment. The model for the 2 time points was considered as an incomplete randomized block model, with each subject as a block, receiving the baseline level in 1 sub-block and either active treatment or placebo in the other sub-block. The generalized estimating equation (GEE) algorithm was used to fit the model, using a robust estimator for the variance which provided a proper adjustment for possible correlation between the 2 measurements on each subject.
  Measure type are estimated mean and measure of dispersion is the standard error of the estimated mean.
Time Frame: Baseline (Days -7 to -1), During Study (Days 1-84)
Population: Full analysis set
Measure: Mean (Standard Error); unit: percentage of total 24 hour periods
Arm/Group | Fp MDPI 12.5 mcg | Fp MDPI 25 mcg | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Placebo MDPI | Flovent Diskus 100mcg
Number analyzed (Participants) | 102 | 101 | 102 | 102 | 102 | 102
percentage of total 24 hour periods | 34.08 (3.909) | 31.76 (4.229) | 28.06 (3.799) | 24.07 (4.283) | 21.30 (4.668) | 29.82 (4.191)
Statistical Analysis 1: Comparison: Fp MDPI 100 mcg vs Placebo MDPI; The generalized estimating equation (GEE) algorithm was used to fit the model, using a robust estimator for the variance which provided a proper adjustment for possible correlation between the 2 measurements on each subject. This model was used to obtain 2-sided 95% confidence limits for the difference in treatment effects of Fp MDPI versus placebo; Test type: Superiority or Other; p = 0.66685, GEE; The model contained covariates for sex, age, and treatment. The baseline level was estimated for all subjects combined, adjusted for covariates; estimated mean difference from placebo = 2.76, 95% CI 2-sided [-10.07 to 15.60]
Statistical Analysis 2: Comparison: Fp MDPI 50 mcg vs Placebo MDPI; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.26741, GEE — The model contained covariates for sex, age, and treatment. The baseline level was estimated for all subjects combined, adjusted for covariates; estimated mean difference from placebo = 6.76, 95% CI 2-sided [-5.43 to 18.94]
Statistical Analysis 3: Comparison: Fp MDPI 25 mcg vs Placebo MDPI; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.09964, GEE — [p-value comment as in outcome 4, analysis 2]; estimated mean difference from placebo = 10.45, 95% CI 2-sided [-2.24 to 23.15]
Statistical Analysis 4: Comparison: Fp MDPI 12.5 mcg vs Placebo MDPI; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.03825, GEE — [p-value comment as in outcome 4, analysis 2]; Slope = 12.78, 95% CI 2-sided [0.44 to 25.11]

5. Secondary Outcome: Kaplan-Meier Estimate of Probability of Remaining in the Study at Week 12
Description: The time to withdrawal due to stopping criteria was compared between the treatment groups with the log rank test. The Kaplan-Meier estimate of the probability of remaining in the study at week 12 with 95% CI was presented by treatment group. Subjects who completed the study were censored at the date of completion, subjects who withdrew for reasons other than stopping criteria were censored at the time of withdrawal. Stopping criteria were based on day subject first met stopping criteria, using subject's diary data and asthma exacerbations recorded in CRF.
Time Frame: Day 1 to Day 84
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Fp MDPI 12.5 mcg | Fp MDPI 25 mcg | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Placebo MDPI | Flovent Diskus 100mcg
Number analyzed (Participants) | 102 | 101 | 102 | 102 | 102 | 102
probability | 0.8041 [0.7067 to 0.8720] | 0.7895 [0.6927 to 0.8589] | 0.9077 [0.8300 to 0.9509] | 0.7657 [0.6660 to 0.8392] | 0.5655 [0.4528 to 0.6636] | 0.8272 [0.7332 to 0.8905]
Statistical Analysis 1: Comparison: Fp MDPI 100 mcg vs Placebo MDPI; Comparison of survival curve to placebo; Test type: Superiority or Other; p = 0.2841, Log Rank — Significance at 0.05
Statistical Analysis 2: Comparison: Fp MDPI 50 mcg vs Placebo MDPI; Comparison of survival curve to placebo; Test type: Superiority or Other; p < 0.0001, Log Rank — Significance at 0.05
Statistical Analysis 3: Comparison: Fp MDPI 25 mcg vs Placebo MDPI; Comparison of survival curve to placebo; Test type: Superiority or Other; p = 0.0008, Log Rank — Significance at 0.05
Statistical Analysis 4: Comparison: Fp MDPI 12.5 mcg vs Placebo MDPI; Comparison of survival curve to placebo; Test type: Superiority or Other; p = 0.0010, Log Rank — Significance at 0.05

6. Secondary Outcome: Area Under The Curve From Time 0 Until The Last Measurable Concentration (AUC0-t) of Fp
Description: Approximately 20% of subjects randomized to the study and distributed across preselected study sites were to participate in fluticasone propionate pharmacokinetic assessments (the pharmacokinetic cohort). Subjects who had received fluticasone propionate in any form (orally, inhaled, or nasal) within 14 days of Day 1 were not permitted to participate in pharmacokinetic assessments.
Time Frame: Day 1: predose (within 10 minutes of treatment administration), and 5, 10, 15, 30, and 45 minutes, 1 hour, 1 hour 15 minutes, 1 hour 30 minutes, and 2, 4, 8, and 12 hours postdose
Population: Pharmacokinetics analysis set. Placebo samples not included in these results.
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | Fp MDPI 12.5 mcg | Fp MDPI 25 mcg | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Placebo MDPI | Flovent Diskus 100mcg
Number analyzed (Participants) | 16 | 22 | 19 | 17 | 0 | 21
pg*hr/mL | 21.6 (27.09) | 42.0 (23.21) | 63.2 (22.64) | 153.8 (91.42) |  | 10.4 (45.65)

7. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Fp
Description: as for outcome 6
Time Frame: as for outcome 6
Population: Pharmacokinetics analysis set. Placebo samples not included in these results.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Fp MDPI 12.5 mcg | Fp MDPI 25 mcg | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Placebo MDPI | Flovent Diskus 100mcg
Number analyzed (Participants) | 16 | 22 | 19 | 17 | 0 | 21
pg/mL | 5.4 (4.23) | 10.0 (5.35) | 12.9 (5.13) | 33.6 (15.49) |  | 23.4 (10.73)

8. Secondary Outcome: Time of Maximum Concentration (Tmax) of Fp
Description: as for outcome 6
Time Frame: as for outcome 6
Population: Pharmacokinetics analysis set. Placebo samples not included in these results.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Fp MDPI 12.5 mcg | Fp MDPI 25 mcg | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Placebo MDPI | Flovent Diskus 100mcg
Number analyzed (Participants) | 16 | 22 | 19 | 17 | 0 | 21
hours | 1.2 (0.97) | 1.4 (2.43) | 1.7 (2.55) | 1.1 (0.95) |  | 1.7 (2.61)

9. Secondary Outcome: Patients With Treatment-Emergent Adverse Experiences (TEAE) During the Treatment Period
Description: An adverse event was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an AE which prevents normal daily activities. Relationship of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Day 1 -84
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Fp MDPI 12.5 mcg | Fp MDPI 25 mcg | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Placebo MDPI | Flovent Diskus 100mcg
Number analyzed (Participants) | 103 | 104 | 104 | 103 | 104 | 104
Participants
  Any adverse event (AE) | 31 | 32 | 36 | 37 | 31 | 32
  Severe AE | 0 | 0 | 3 | 2 | 3 | 3
  Treatment-related AE | 6 | 3 | 3 | 2 | 1 | 1
  Deaths | 0 | 0 | 0 | 0 | 0 | 0
  Other serious AE | 0 | 0 | 1 | 2 | 2 | 2
  Withdrawn from treatment due to AE | 0 | 0 | 0 | 1 | 2 | 2

10. Secondary Outcome: Oropharyngeal Exam Findings at Each Study Visit
Description: Oropharyngeal examinations for visual evidence of oral candidiasis were conducted at all study visits. If the visual oropharyngeal examination was abnormal at the screening visit, the subject was excluded from entering the study and subjects with an abnormal oropharyngeal exam on Day 1 were not eligible for randomization. Any visual evidence of oral candidiasis during the treatment period of the study was evaluated by obtaining and analyzing a swab of the suspect area. Appropriate therapy was to be initiated immediately at the discretion of the investigator and was not to be delayed for culture confirmation. Subjects with a culture-positive infection could continue participation in the study on appropriate anti-infective therapy, provided this therapy was not prohibited by the protocol. If a subject required a protocol-prohibited medication for therapy, the subject was to be discontinued from the study.
  Data format: Time frame, <signs of oral candidiasis?> yes or no
Time Frame: Screening (week -3 to -2), Baseline (Week 0), Weeks 1, 2, 4, 8, 12
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Fp MDPI 12.5 mcg | Fp MDPI 25 mcg | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Placebo MDPI | Flovent Diskus 100mcg
Number analyzed (Participants) | 103 | 104 | 104 | 103 | 104 | 104
Participants
  Screening - Yes: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Screening - Yes | 0 | 0 | 0 | 0 | 0 | 0
  Screening - No | 103 | 104 | 104 | 103 | 104 | 104
  Week 0 - Yes: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Week 0 - Yes | 0 | 0 | 0 | 0 | 0 | 0
  Week 0 - No | 103 | 104 | 104 | 103 | 104 | 104
  Week 1 - Yes: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Week 1 - Yes | 0 | 0 | 0 | 0 | 0 | 0
  Week 1 - No: number analyzed (Participants) | 93 | 98 | 100 | 100 | 94 | 98
  Week 1 - No | 93 | 98 | 100 | 100 | 94 | 98
  Week 2 - Yes: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Week 2 - Yes | 0 | 0 | 0 | 0 | 0 | 0
  Week 2 - No: number analyzed (Participants) | 90 | 93 | 99 | 95 | 83 | 93
  Week 2 - No | 90 | 93 | 99 | 95 | 83 | 93
  Week 4 - Yes (positive culture): number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Week 4 - Yes (positive culture) | 0 | 1 | 0 | 0 | 0 | 0
  Week 4 - No: number analyzed (Participants) | 88 | 89 | 97 | 91 | 75 | 90
  Week 4 - No | 88 | 89 | 97 | 91 | 75 | 90
  Week 8 - Yes: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 - Yes | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 - No: number analyzed (Participants) | 84 | 85 | 92 | 84 | 66 | 83
  Week 8 - No | 84 | 85 | 92 | 84 | 66 | 83
  Week 12 - Yes: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Week 12 - Yes | 0 | 0 | 0 | 0 | 0 | 0
  Week 12 - No: number analyzed (Participants) | 102 | 102 | 103 | 100 | 97 | 101
  Week 12 - No | 102 | 102 | 103 | 100 | 97 | 101

11. Other Pre Specified Outcome: Change From Baseline In Trough (Morning Predose And Pre-Rescue Bronchodilator) Forced Expiratory Volume In 1 Second (FEV1) Over The 12-Week Treatment Period Inclusive of Flovent Diskus Data
Description: Trough FEV1 was measured electronically by spirometry at morning (AM) investigational site visits, before administration of the AM dose of study drug and before albuterol/salbutamol administration. The highest FEV1 value from 3 acceptable and 2 reproducible maneuvers was used. All FEV1 data were submitted to a central reading center for evaluation.
  The p-values for the treatment comparisons to placebo are from an MMRM model including data from all treatments: change from baseline = baseline FEV1 + sex + age + treatment + visit + treatment*visit with an unstructured covariance matrix assumed.
Time Frame: Baseline (Day 1, pre-dose), During Study (Days 7, 14, 28, 56 and 84 pre-dose)
Population: Full analysis set, (participants who contributed >=1 to the analysis). Data from one site omitted due to GCP concerns.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Fp MDPI 12.5 mcg | Fp MDPI 25 mcg | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Placebo MDPI | Flovent Diskus 100mcg
Number analyzed (Participants) | 94 | 97 | 100 | 94 | 94 | 96
liters | 0.172 (0.0293) | 0.232 (0.0288) | 0.245 (0.0280) | 0.268 (0.0292) | 0.120 (0.0294) | 0.234 (0.0288)
Statistical Analysis 1: Comparison: Placebo MDPI vs Flovent Diskus 100mcg; Test type: Superiority or Other; p = 0.0058, mixed model for repeated measures — Significance at 0.05; LSM difference = -0.114, 95% CI 2-sided [-0.195 to -0.033]
Statistical Analysis 2: Comparison: Fp MDPI 100 mcg vs Flovent Diskus 100mcg; Test type: Superiority or Other; p = 0.4083, mixed model for repeated measures — Significance at 0.05; LSM difference = 0.034, 95% CI 2-sided [-0.046 to 0.114]
Statistical Analysis 3: Comparison: Fp MDPI 50 mcg vs Flovent Diskus 100mcg; Test type: Superiority or Other; p = 0.7882, mixed model for repeated measures — Significance at 0.05; LSM difference = 0.011, 95% CI 2-sided [-0.068 to 0.089]
Statistical Analysis 4: Comparison: Fp MDPI 25 mcg vs Flovent Diskus 100mcg; Test type: Superiority or Other; p = 0.9586, mixed model for repeated measures — Significance at 0.05; LSM difference = -0.002, 95% CI 2-sided [-0.082 to 0.078]
Statistical Analysis 5: Comparison: Fp MDPI 12.5 mcg vs Flovent Diskus 100mcg; Test type: Superiority or Other; p = 0.1306, mixed model for repeated measures — Significance at 0.05; LSM difference = -0.062, 95% CI 2-sided [-0.143 to 0.018]

12. Other Pre Specified Outcome: Change From Baseline In Weekly Average Of Daily Trough (Predose And Pre-Rescue Bronchodilator) Morning Peak Expiratory Flow (PEF) Over The 12-Week Treatment Period Inclusive of Flovent Diskus Data
Description: Peak expiratory flow was determined in the AM and in the PM, before administration of study or rescue medications using a handheld electronic peak flow meter. The highest value of triplicate measurements obtained was recorded by the subject's diary device.
  On mornings for which a treatment visit was scheduled (TV1 through TV9), the PEF was measured and recorded at the investigational site visit.
  Baseline trough AM PEF was defined as the average of recorded (non-missing) trough AM PEF assessments over the 7 days directly preceding first study drug intake.
  The p-values for the treatment comparisons to placebo are from an MMRM model including all treatments: change from baseline = baseline PEF + sex + age + treatment + visit + treatment*visit with an unstructured covariance matrix assumed.
Time Frame: Baseline (Days -7 to 1, am pre-dose), During Study (Days 2-84 am pre-dose)
Population: Full analysis set, (participants who contributed >=1 to the analysis). Data from one site omitted due to GCP concerns.
Measure: Least Squares Mean (Standard Error); unit: liters/minute
Arm/Group | Fp MDPI 12.5 mcg | Fp MDPI 25 mcg | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Placebo MDPI | Flovent Diskus 100mcg
Number analyzed (Participants) | 94 | 97 | 99 | 94 | 92 | 96
liters/minute | 31.20 (4.544) | 21.27 (4.465) | 29.63 (4.339) | 27.66 (4.550) | 9.30 (4.700) | 26.96 (4.496)
Statistical Analysis 1: Comparison: Placebo MDPI vs Flovent Diskus 100mcg; Test type: Superiority or Other; p = 0.0068, mixed model for repeated measures — Significance at 0.05; LSM difference = -17.66, 95% CI 2-sided [-30.43 to -4.89]
Statistical Analysis 2: Comparison: Fp MDPI 100 mcg vs Flovent Diskus 100mcg; Test type: Superiority or Other; p = 0.9135, mixed model for repeated measures — Significance at 0.05; LSM difference = 0.69, 95% CI 2-sided [-11.84 to 13.23]
Statistical Analysis 3: Comparison: Fp MDPI 50 mcg vs Flovent Diskus 100mcg; Test type: Superiority or Other; p = 0.6689, mixed model for repeated measures — Significance at 0.05; LSM difference = 2.67, 95% CI 2-sided [-9.58 to 14.92]
Statistical Analysis 4: Comparison: Fp MDPI 25 mcg vs Flovent Diskus 100mcg; Test type: Superiority or Other; p = 0.3691, mixed model for repeated measures — Significance at 0.05; LSM difference = -5.69, 95% CI 2-sided [-18.12 to 6.74]
Statistical Analysis 5: Comparison: Fp MDPI 12.5 mcg vs Flovent Diskus 100mcg; Test type: Superiority or Other; p = 0.5072, mixed model for repeated measures — Significance at 0.05; LSM difference = 4.24, 95% CI 2-sided [-8.31 to 16.78]

13. Other Pre Specified Outcome: Change From Baseline In Weekly Average Of Daily Evening Peak Expiratory Flow (PEF) Over The 12-Week Treatment Period Inclusive of Flovent Diskus Data
Description: Peak expiratory flow was determined in the AM and in the PM, before administration of study or rescue medications using a handheld electronic peak flow meter. The highest value of triplicate measurements obtained was recorded by the subject's diary device.
  PM PEF baseline was defined as the average of recorded (nonmissing) PM PEF assessments over the 7 days directly preceding first study drug intake.
  The p-values for the treatment comparisons to placebo are from an MMRM model including all treatment groups: change from baseline = baseline PEF + sex + age + treatment + visit + treatment*visit with an unstructured covariance matrix assumed.
Time Frame: Baseline (Days -7 to 1, am pre-dose), During Study (Days 2-84 am pre-dose)
Population: Full analysis set, (participants who contributed >=1 to the analysis). Data from one site omitted due to GCP concerns.
Measure: Least Squares Mean (Standard Error); unit: liters/minute
Arm/Group | Fp MDPI 12.5 mcg | Fp MDPI 25 mcg | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Placebo MDPI | Flovent Diskus 100mcg
Number analyzed (Participants) | 92 | 98 | 99 | 92 | 92 | 95
liters/minute | 28.00 (4.442) | 18.97 (4.315) | 22.27 (4.206) | 20.47 (4.453) | 9.70 (4.557) | 24.95 (4.356)
Statistical Analysis 1: Comparison: Placebo MDPI vs Flovent Diskus 100mcg; Test type: Superiority or Other; p = 0.0158, mixed model for repeated measures — Significance at 0.05; LSM difference = -15.26, 95% CI 2-sided [-27.63 to -2.88]
Statistical Analysis 2: Comparison: Fp MDPI 100 mcg vs Flovent Diskus 100mcg; Test type: Superiority or Other; p = 0.4709, mixed model for repeated measures — Significance at 0.05; LSM difference = -4.48, 95% CI 2-sided [-16.69 to 7.721]
Statistical Analysis 3: Comparison: Fp MDPI 50 mcg vs Flovent Diskus 100mcg; Test type: Superiority or Other; p = 0.6572, mixed model for repeated measures — Significance at 0.05; LSM difference = -2.68, 95% CI 2-sided [-14.55 to 9.19]
Statistical Analysis 4: Comparison: Fp MDPI 25 mcg vs Flovent Diskus 100mcg; Test type: Superiority or Other; p = 0.3292, mixed model for repeated measures — Significance at 0.05; LSM difference = -5.98, 95% CI 2-sided [-18.01 to 6.05]
Statistical Analysis 5: Comparison: Fp MDPI 12.5 mcg vs Flovent Diskus 100mcg; Test type: Superiority or Other; p = 0.6237, mixed model for repeated measures — Significance at 0.05; LSM difference = 3.05, 95% CI 2-sided [-9.16 to 15.26]

ADVERSE EVENTS:
Time Frame: Day 1 to 84
Groups:
- Flovent Diskus 100mcg: Fluticasone propionate (Fp) 100 mcg per dose twice a day (for a total daily dose of 200 mcg) using a multidose dry powder inhaler (MDPI) for 12 weeks in an open-label manner.
- Fp MDPI 100 mcg: Fluticasone propionate (Fp) 100 mcg per dose twice a day (for a total daily dose of 200 mcg) using a multidose dry powder inhaler (MDPI) for 12 weeks in a double-blind manner.
- Fp MDPI 12.5 mcg: Fluticasone propionate (Fp) 12.5 mcg per dose twice a day (for a total daily dose of 25 mcg) using a multidose dry powder inhaler (MDPI) for 12 weeks in a double-blind manner.
- Fp MDPI 25 mcg: Fluticasone propionate (Fp) 25 mcg per dose twice a day (for a total daily dose of 50 mcg) using a multidose dry powder inhaler (MDPI) for 12 weeks in a double-blind manner.
- Fp MDPI 50 mcg: Fluticasone propionate (Fp) 50 mcg per dose twice a day (for a total daily dose of 100 mcg) using a multidose dry powder inhaler (MDPI) for 12 weeks in a double-blind manner.
- Placebo MDPI: Placebo twice a day using a multidose dry powder inhaler (MDPI) for 12 weeks in a double-blind manner.
Arm/Group | Flovent Diskus 100mcg | Fp MDPI 100 mcg | Fp MDPI 12.5 mcg | Fp MDPI 25 mcg | Fp MDPI 50 mcg | Placebo MDPI
Serious Adverse Events (participants affected / at risk) | 2/104 | 2/103 | 0/103 | 0/104 | 1/104 | 2/104
Other Adverse Events (participants affected / at risk) | 5/104 | 8/103 | 10/103 | 7/104 | 10/104 | 8/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flovent Diskus 100mcg (N=104) | Fp MDPI 100 mcg (N=103) | Fp MDPI 12.5 mcg (N=103) | Fp MDPI 25 mcg (N=104) | Fp MDPI 50 mcg (N=104) | Placebo MDPI (N=104)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flovent Diskus 100mcg (N=104) | Fp MDPI 100 mcg (N=103) | Fp MDPI 12.5 mcg (N=103) | Fp MDPI 25 mcg (N=104) | Fp MDPI 50 mcg (N=104) | Placebo MDPI (N=104)
Nasopharyngitis (Infections and infestations) | 1 (3) | 3 (3) | 4 (4) | 5 (5) | 7 (7) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 5 (5) | 7 (7) | 2 (2) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.